CLINICAL TRIAL: NCT04962256
Title: The Application of Enhanced Recovery After Surgery (ERAS) During the Perioperative Period of Patients With Posterior Approach of Cervical Spine Operation: a Mixed Methods Study
Brief Title: ERAS in Posterior Approach of Cervical Spine Operation
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019144
Record Dates: First submitted 2021-06-27; First posted 2021-07-14 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Cervical Myelopathy
Keywords: Cervical Myelopathy; Enhanced recovery after surgery; Surgical outcome
MeSH Terms: interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients with degenerative CSM or OPLL undergoing C3-7 open-door laminoplasty
  Interventions: Procedure: Enhanced recovery after surgery

INTERVENTIONS:
Procedure: Enhanced recovery after surgery — ERAS management includes 3 parts: (1) Preoperative analgesia and airway evaluation. (2) The protection and reconstruction of the musculo-ligamentous complex during the surgery, the safe intubation, and the local infiltration anesthesia during surgery. (3) Collar free, multimodal analgesia, airway management, and early recovery after surgery.

SUMMARY:
Enhanced recovery after surgery (ERAS) strategy has been used in the patient management of different diseases. This study aims to evaluate the effectiveness of ERAS in the perioperative period of posterior approach of cervical spine operation among patients with CSM.

DETAILED DESCRIPTION:
Enhanced recovery after surgery (ERAS) strategy has been used in the patient management of different diseases, but up to now, few effort has been done to evaluate the effectiveness of ERAS in patients perioperative management of cervical spine surgery. As a interdisciplinary cooperation system, either qualitative or quantitative method alone can not completely reflect the function of ERAS. Mixed model research (MMR) is a appropriate method to evaluate a complex system, but it has not been used in ERAS evaluation. This study aims to evaluate the effectiveness of ERAS in the perioperative period of posterior approach of cervical spine operation among patients with CSM using MMR, including the retrospective quantitative part and prospective qualitative part. In the retrospective part, we will collect the data of length of stay, VAS scores, mJOA scores and SF-36 scores to compare the difference between ERAS group and regular group. In the prospective part, we will collect the data from the focus group meetings and personal interviews of patients, to verify that ERAS has the ability to improve the postoperative outcomes, while maintain an equal surgical effect.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should be diagnosed as CSM based on the history, symptoms, Physical signs and radiographic results.
2. Patients did not respond to the 3-month conventional treatment.
3. Patients were performed posterior approach of cervical spine operation.
4. Patients should have complete pre- and post-operative data.

Exclusion Criteria:

1. Patients with severe organic diseases.
2. Patients with previous history of cervical spine surgery.
3. Patients with mental or psychological abnormality.
4. Patients with severe osteoporosis (T value <-2.5).

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with posterior approach of cervical spine operation
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Outcomes of pain | Preoperation
  Visual analogue scale before after surgery, 0 to 10 points, higher means severer the pain is.
Outcomes of pain | 3 months after surgery.
  Visual analogue scale 3-month after surgery, 0 to 10 points, higher means severer the pain is.
Length of stay | Admission to discharge, an average of 3 days
  Length of stay
Neurological function | Preoperation
  Modified Japanese Orthopaedic Association score before surgery, -2 to 17 points, higher means better outcome.
Neurological function | 3 months after surgery.
  Modified Japanese Orthopaedic Association score 3-month after surgery, -2 to 17 points, higher means better outcome.
Outcomes of quality of life | Preoperation
  36-Item Short Form Survey score before surgery, 0 to 100 points, higher means better outcome.
Outcomes of quality of life | 3 months after surgery
  36-Item Short Form Survey score 3-month after surgery, 0 to 100 points, higher means better outcome.
Focus group meetings | Admission to discharge, an average of 3 days
  Focus group meetings by specialists, to discuss the effect of ERAS and the what improvements can be made.
Personal interviews | At 3-month follow-up
  Personal interviews of patients at 3-month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Feifei Zhou, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No